CLINICAL TRIAL: NCT01206751
Title: Multi-detector Computer Tomography Protocol Project: Chest Imaging Technique and Case Presentation
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wing P. Chan, Wan Fang Hospital Department of Radiology
Other Study IDs: 99008
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Aortic Dissection; Thrombosis in Left Atrium and Right Axillary Artery; Double IVC; May-Thurner Syndrome; Pulmonary Thromboembolism
MeSH Terms: conditions — Aortic Dissection; May-Thurner Syndrome; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Chest imaging technique and case presentation

SUMMARY:
Multi-detector computer tomography protocol project: Chest imaging technique and case presentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete clinical images

Exclusion Criteria:

* Patients with incomplete clinical images

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with complete clinical images
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wing P. Chan, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan